CLINICAL TRIAL: NCT04078204
Title: A Multi-center, Randomized, Double-Blind, Placebo-Controlled Study of Dl-3-Butylphthalide on the Treatment of Small Cerebral Vessel Disease
Brief Title: A Clinical Study on the Treatment of Cerebral Small Vascular Disease
Acronym: MAP-CSVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018ZX09711001-003-021
Record Dates: First submitted 2019-02-24; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: Butylphthalide; Cerebral Small Vessel Diseases; Clinical Study
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butylphthalide Soft Capsules (Experimental): Two Butylphthalide soft capsules will be taken three times a day before meals.
  Interventions: Drug: Butylphthalide Soft Capsules
- Placebo Soft Capsules (Placebo Comparator): Two placebo soft capsules will be taken three times a day before meals.
  Interventions: Drug: placebo Soft Capsules

INTERVENTIONS:
Drug: Butylphthalide Soft Capsules — The experimental group will receive the Butylphthalide Soft Capsules during the 24-month intervention period. After the 24-month intervention,The experimental group will receive Butylphthalide Soft Capsules for the 6-month open treatment period.
  Arms: Butylphthalide Soft Capsules
Drug: placebo Soft Capsules — The placebo group will receive the Placebo Soft Capsules during the 24-month intervention period. After the 24-month intervention,The placebo group will receive Butylphthalide Soft Capsules for the 6-month open treatment period.
  Arms: Placebo Soft Capsules

SUMMARY:
This study is designed to evaluate the safety and efficacy of butylphthalide (NBP) in the treatment of cerebral small vessel disease through a multicenter, randomized,double-blind, placebo-controlled study. Butylphthalide Soft Capsule and placebo were prescribed to the experimental group and the control group for a period of 24-months, respectively. After that, the experimental group and the control group were given Butylphthalide Soft Capsule for 6 months.

DETAILED DESCRIPTION:
Butylphthalide can protect mitochondrial function and inhibit neuronal apoptosis by significantly increasing the activity of mitochondrial ATP complex enzyme and mitochondrial respiratory chain complex enzyme IV, improving the fluidity of mitochondrial membrane and maintaining mitochondrial membrane potential. Butylphthalide can reconstruct microcirculation and protect mitochondria, which can protect neurovascular units in an all-round way. Findings from previous studies have shown that butylphthalide can improve the ability of daily living of patients with ischemic cerebrovascular disease and can enhance cognitive function of patients diagnosed as subcortical vascular cognitive impairment no dementia.

ELIGIBILITY:
Inclusion Criteria:

1. 50-80 years of age;
2. all subjects with a culture level of primary school or above;
3. Cerebral MRI demonstrated that patients with white matter hyperintense signal of vascular origin (Fazekas score≥ 2 points) and lacunar lesions (≥ 2);
4. Consistent with at least one of the following clinical manifestations: (1)Subjects with a history of lacunar stroke syndrome more than 6-months before study initiation(Patients should have one of the traditional clinical lacunar syndromes and a new symptomatic lesion with a diameter of less than 20mm observed in subcortical white matter or basal ganglia), without a stenosis of greater than 50% in ipsilateral internal carotid artery or middle cerebral artery.) (2)Subjects with cognitive impairment (impairment involving memory and/or other cognitive domains and lasting for at least 3-months) have at least one domain rating of CDR > 0.5. Cognitive impairment and cerebrovascular disease are likely to have a causal relationship, showing sudden or fluctuating cognitive decline with ladder-like progress.
5. Modified Rankin score ≤ 3 points; MMSE ≥ 10 points;
6. Subjects have stable and reliable caregivers who must be able to communicate frequently with the subjects (at least 4 days a week, at least 2 hours a day). The caregivers will help the subjects participate in the whole process of the study. The caregiver must accompany the subjects to participate in the research visits, and must fully interact and communicate with the subjects in order to provide valuable information for CIBIC-plus, ADL, NPI and other scales.
7. Female patients are menopausal women (menopause ≥ 24 weeks), or have undergone surgical sterilization or have agreed to take effective contraceptive measures during the trial period.
8. If patients use antipsychotic drugs (risperidone, quetiapine or olanzapine), anti-anxiety and depression drugs, sedative and hypnotic drugs and other drugs before screening, they need to take them stably for at least one month before screening, and try to maintain the dose stability during the research process. Sedative and hypnotic drugs such as zopiclone, alprazolam and estazolam may be used when necessary, but they should not be used within 8 hours of visiting time.
9. Consent to participation in this study with the written informed consents obtained from all patients or their legal surrogates.

Exclusion Criteria:

1. New onset cerebral infarction or intracranial hemorrhage within 6 months;
2. Complicated with cerebral cortical infarction or cerebral hemorrhage,hydrocephalus and other white matter lesions of non-vascular origin (multiple sclerosis, carbon monoxide poisoning encephalopathy, etc.);
3. Systemic diseases that may be responsible for cognitive impairment (such as liver and kidney dysfunction, endocrine diseases, vitamin deficiency, systemic autoimmune diseases, etc.);
4. Depression and depression related conditions (Hamilton Depression Scale score ≥ 17 points), or other unrelated serious mental disorders (schizophrenia, bipolar affective disorder or delirium) or serious neurological diseases (such as central nervous system infection (for example AIDS, syphilis), Creutzfeldt-Jakob disease, Huntington's chorea and primary Parkinson's disease,Lewy body dementia,corticobasal ganglia degeneration, brain trauma, epilepsy, brain tumors (with an exception of patients with meningioma which could not attribute to cognitive impairment based on the judgement of the researchers.)
5. Those who use other drugs that affect the safety or efficacy evaluation of the tested drugs and disagree with withdrawal, such as NBP,cholinesterase inhibitors (Arizona, Essene, Galantamine, Huperzine A Tablets, Benzhexol Hydrochloride etc.), N-methyl-D-aspartic acid (NMDA) antagonists (such as Memantine, Amantadine, Ketamine, etc.);
6. Patients allergic or intolerant to butylphthalide (NBP) ;
7. Patients with severe cardiac,pulmonary and renal insufficiency (creatinine > 2.0 mg/dl or 178umol/L), severe liver dysfunction (ALT or AST >3 times of upper limit of the normal value), any malignancies and those with a life expectancy less than 2 years;
8. Patients with Coagulation dysfunction or thrombocytopenia (platelet < 100 *10^9/L);
9. Contraindication for MR examination.
10. Women during pregnancy and lactation period or plan to be pregnant.
11. Patients who are participating in other interventional clinical studies or have participated in other interventional clinical studies in the past three months;
12. Patients who could not be followed up as required during the study period;
13. Patients unable to complete neuropsychological evaluations due to illiteracy or irreparable audiovisual impairment;
14. Refractory hypertension: blood pressure ≥180/110 mmHg;
15. The subjects are the investigators and immediate family members participating in the study, employees and immediate family members of embip.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The occurrence of the composite endpoint | 30 months
  new stroke event (ischemic or haemorrhagic), new onset dementia, an increase of modified Rankin Score (mRS) by ≥2 points, severe disability (mRS≥5), or death
Change of CIBIC-Plus score | 30 months
  Through interviews with caregivers and patients, a brief assessment of the patient's mental state was made in terms of the patient's relevant history, physical appearance, psychological/cognitive status, behavior, and ability to live daily. According to the above, the patients were evaluated: 1) significant improvement, 2) improved vector, 3) slight improvement, 4) no change, 5) slight deterioration, 6) moderate deterioration, and 7) severe deterioration.
Change of ADAS-cog score | 30 months
  1. Recall common words
  2. Name the 12 objects submitted and the fingers on the hand
  3. Understand and complete 1-5 steps
  4. Copy 4 geometric shapes
  5. The ability to complete familiar but complex sequence activities
  6. Evaluation of time and place orientation
  7. Identify new words from words already given
  8. Remember the instructions in the cognitive task
  9. Evaluation of patients' ability to speak and communicate
  10. Evaluation of patients' language ability
  11. Ability to understand spoken language
  12. Patient attention during measurement Scoring criteria for (1)-(7) :The score is incorrect number of steps. Scoring criteria for (8)-(12) : 0= none, 1= very light, 2= mild, 3= moderate, 4= moderate, 5= severe.
Volume changes of white matter hyperintensities observed on cerebral MRI | 30 months
  Nothing

SECONDARY OUTCOMES:
The proportion of participants with an increase of mRS by≥ 2, or mRS≥5 for severe disability | 30 months
  Level 1: symptomatic, but not obviously disabled, able to complete daily work and activities Level 2: mildly disabled, unable to complete daily activities before illness, but able to take care of themselves Level 3: moderately disabled, needs some help, but cannot walk without help Level 4: moderate to severe disability, need help walking, need help to complete their own care Level 5: severely disabled, bedridden, incontinence, need daily care Level 6: death
The proportion of participants with new onset dementia。New onset dementia meets the following three criteria: | 30 months
  1. Mini-Mental State Examination (MMSE) score<20 (primary school) or < 24 points (junior high school or above); MMSE is a scale assessing orientation, memory, attention, language, and visuospatial function. Scores in each item are combined to obtain a total score ranging from 0 to 30. Score of 24 or more indicates normal cognition
  2. Clinical Dementia Rating-Sum of Boxes (CDR-SB)≥1 CDR assesses cognitive performance in six areas: memory, orientation, judgment & problem solving, community affairs, home & hobbies, and personal care. Scores in each of these are combined to obtain a composite score ranging from 0 to 3
  3. Instrumental Activities of Daily Living (IADLs)>26 points IADLs scale assesses 20 items of daily living ability. The score of each item ranges from 1 to 4 points: 1 is normal, and 4 indicate obvious functional decline. Scores in each item are combined to obtain a total score ranging from 20 to 80
The proportion of participants with death due to any known or unknown cause | 30 months
  The causes of death were classified as follows: ischemic stroke, hemorrhagic stroke, heart disease , hemorrhage (excluding intracranial hemorrhage), infection, malignant tumors, trauma, other vascular etiology (including pulmonary embolism), other non-vascular and unclear etiology.
Changes of the gait speed in three-meter walktest | 30 months
  Nothing
Changes in the number of silent brain infarcts | 30 months
  Nothing
Changes in the number of cerebral microbleeds | 30 months
  Nothing
Evolution of brain volumes (gray matter, white matter and CSF volumes) | 30 months
  Nothing

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided